CLINICAL TRIAL: NCT06107595
Title: A Randomized Controlled Trial Evaluating the Efficacy of Conditioned Open Label Placebo (COLP) to Limit Opioid Reliance for Postoperative Pain Management
Brief Title: Conditioned Open Label Placebo for Postoperative Pain Management
Acronym: COLP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre de Médecine Intégrative et Complémentaire (CEMIC) (Other)
Responsible Party: Principal Investigator, Chantal Berna Renella, Professor, Centre de Médecine Intégrative et Complémentaire (CEMIC)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-01664
Record Dates: First submitted 2023-10-18; First posted 2023-10-30 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Efficacy of conditioned open label placebo pill (Experimental): On postoperative day 0, participant will self-administer one OLP with all opioid analgesics (whether administered intravenously or orally). This pairing will be done from postoperative day 0 to postoperative day 17.
  Starting on postoperative day 2, participants take 3 scheduled placebo doses (pills or inhalation) every day, at 3 convenient times. In parallel, the OLP pairing to standard and rescue doses of opioids will continue.
  The patients are told to continue taking both scheduled standalone COLP and paired COLP (if needed) until postoperative day 17.
  Interventions: Behavioral: Placebo
- Efficacy of conditioned open label placebo odor (Experimental): 1 drops of clove oil (i.e. eugenol) will be disposed on a cotton and inserted into a stick. The patients will be asked to actively smell them by sniffing using a stick of inhalation. On postoperative day 0, participant will self-administer one OLP with all opioid analgesics (whether administered intravenously or orally). This pairing will be done from postoperative day 0 to postoperative day 17.
  On postoperative day 2, participants take 3 scheduled placebo doses (pills or inhalation) every day, at 3 convenient times. In parallel, the OLP pairing to standard and rescue doses of opioids will continue.
  The patients are told to continue taking both scheduled standalone COLP and paired COLP (if needed) until postoperative day 17
  Interventions: Behavioral: Placebo
- Standard of care (Active Comparator): Usual postoperative pain management, relying mainly on opioids
  Interventions: Behavioral: Placebo

INTERVENTIONS:
Behavioral: Placebo — Participant take 1 dose placebo (odor or pill) on post-op day 0 (POD 0) and 3 placebo dose from POD 2 to POD 17

SUMMARY:
The primary objective is to evaluate the efficacy of two Conditioned Open Label Placebos (COLP): COLP pill and COLP odor to reduce opioid intake for postoperative (thoracic and spinal surgery) pain management compared to the opioid only usual treatment (TAU).

DETAILED DESCRIPTION:
Patients, eligible for an elective thoracic or spinal surgery, will be randomized into either standard of care, COLP_pill or COLP_odor. Patients in COLP groups will be asked to pair each opioid intake with an open label placebo intake (either a pill or an inhalation) for postoperative (POD) day 0 to 17. From POD 2, patients in the intervention arms will be additionally asked to take OLP alone 3 times a day. Patients will have unrestricted access to pain killers. Patients will daily assess opioid intake, pain intensity, side effects, mobility and sense of agency using a e-dairy.

ELIGIBILITY:
Inclusion Criteria:

* Spinal or thoracic elective surgery for the indications mentioned above
* Able to give informed consent
* Interested in trying COLP as complementary pain management therapy
* Able to fill a e-diary at home

Exclusion Criteria:

* Cognitive impairment (MOCA score <26)
* Inability to engage in the intervention of the study e.g. inability to communicate in French without a translator, severe hearing impairment without any hearing aid available at the time of intervention, anosmia or intolerance to eugenol.
* Acute psychiatric (e.g. psychotic or suicidal ideation) or somatic (e.g. unstable cardio-respiratory condition) co-morbidity preventing full engagement during intervention
* Opioid use disorder (toxicomania) or contraindication to pain management using opioids (allergy, refusal, ...)
* Intolerance to placebo ingredients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Opioids consumption | 17 days
  Cumulative opioids intake as postoperative consumption (in MgMeq)

SECONDARY OUTCOMES:
Time to Opioid withdrawal (in days) | until the 6 months follow-up
  Time to Opioid withdrawal calculated for COLP compared to treatment as usual
Postoperative pain intensity | 17 days
  Daily Visual Analog Score from the e-diary (score from 0 to 10, 10=worst pain)
Satisfaction with postoperative management | 17 days
  Daily Visual Analog Score from the e-diary (score from 0 to 10, 10=highest satisfaction)
Mobility | 17 days
  Daily Visual Analog Score from the e-diary (score from 0 to 10, 10=best ability to move)
Sense of agency | 17 days
  Daily Visual Analog Score from the e-diary (score from 0 to 10, 10=best sense of agency)
Side effects intensity | 17 days
  Daily Visual Analog Score from the e-diary (score from 0 to 10, 10=worst intensity)

CONTACTS AND LOCATIONS:
Overall Officials: Chantal Berna Renella, Prof, Principal Investigator — Centre de Médecine Intégrative et Complémentaire, Lausanne University hospital
Locations (1):
- Centre de Médecine Intégrative et Complémentaire, Service d'anesthésiologie, CHUV,, Lausanne, Canton of Vaud, Switzerland